CLINICAL TRIAL: NCT01675596
Title: A Multicentre, Non-Randomised Controlled Study of the Safety, Performance, Quality of Life and Cost Effectiveness Outcomes of the Edwards SAPIEN XT™ Transcatheter Heart Valve in an Australian Population
Brief Title: The SOLACE-AU Clinical Trial
Acronym: SOLACE-AU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Collaborators: Pacific Clinical Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-14
Record Dates: First submitted 2012-08-28; First posted 2012-08-30 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-03

CONDITIONS: Severe, Symptomatic Aortic Stenosis
Keywords: Aortic Stenosis; Transfemoral; Transcatheter Heart Valve
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Test (Experimental): SAPIEN XT™ valve with the NovaFlex and NovaFlex+ delivery systems.
  Interventions: Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis

INTERVENTIONS:
Device: TAVR Implantation of the Transcatheter Aortic Valve Prosthesis — Operable subjects
  Other Names: Implantation of the Transcatheter Aortic Valve Prosthesis

SUMMARY:
The objective of the study is to observe the safety, efficacy and cost effectiveness of the Edwards SAPIEN XT valve for the treatment of severe calcific degenerative aortic stenosis.

DETAILED DESCRIPTION:
This is a multi-centre, prospective, consecutively enrolled, non-randomized clinical trial. The comparatator group will consist of subjects undergoing surgical aortic valve replacement in Cohort A of the PARTNER II Trial [NCT01314313].

ELIGIBILITY:
Inclusion Criteria:

* Age > 70 years
* STS Score > 4
* Heart team agrees on eligibility including assessment that TAVR or AVR is appropriate

Exclusion Criteria:

* Age <70 years
* Evidence of an acute myocardial infarction ≤ 30 days
* Aortic valve is a congenital unicuspid or congenital bicuspid valve, or is non-calcified
* Stroke or transient ischemic attack (TIA) within 6 months of the procedure

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 199 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Owen Christopher Raffel, Principal Investigator — The Prince Charles Hospital
Locations (11):
- Australia (11):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - Macquarie Unversity Hospital, Macquarie Park, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - The Prince Charles Hospital, Chermside, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - The Alfred Hospital, Melbourne, Victoria
  - St Vincent's Hospital - MELBOURNE, Melbourne, Victoria
  - Royal Melbourne Hospital, Parkville, Victoria
  - Royal Perth Hospital/Fiona Stanley Hospital, Perth, Western Australia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- TAVR With SAPIEN XT THV: SAPIEN XT™ THV with the NovaFlex and NovaFlex+ delivery systems.
  TAVR Implantation of the Transcatheter Aortic Valve Prosthesis: Operable subjects
Period: Overall Study
Arm/Group | TAVR With SAPIEN XT THV
Started | 199 (One patient did not receive the study device.)
Completed (30 day follow-up) | 191
Not Completed | 8
Not completed — Death | 6
Not completed — Exit with other reason | 1
Not completed — Missed Visit | 1

BASELINE CHARACTERISTICS:
Arm/Group | TAVR With SAPIEN XT THV
Number analyzed (Participants) | 199
Age, Continuous [Mean (Standard Deviation); unit: Years] | 85.5 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108
  Male | 91
STS Score [Mean (Standard Deviation); unit: units on a scale] — The Society of Thoracic Surgeons (STS) score measures patient risk at the time of cardiovascular surgery on a scale that ranges from 0% to 100%, with higher numbers indicating greater risk.
  units on a scale | 5.9 (2.59)
NYHA I/II [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  Participants | 43
NYHA III/IV [Count of Participants; unit: Participants] — New York Heart Association (NYHA), functional classification of heart failure based on how much a patient is limited during physical activity. The rating ranges from I - IV, with the lowest as no limitations and the highest unable to carry on any physical activity without discomfort.
  Participants | 156

OUTCOME MEASURES:

1. Primary Outcome: VARC-2 Composite Safety Endpoint
Description: The primary endpoint is a VARC-2 Composite. It comprises of
  1. All cause mortality
  2. All stroke
  3. Life-threatening bleeding
  4. Acute kidney injury - Stage 3 (including renal replacement therapy)
  5. Coronary artery obstruction requiring intervention
  6. Major vascular complications
  7. Valve related dysfunction (requiring repeat procedure)
  A composite endpoint is an endpoint that is a combination of multiple components.
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | TAVR With SAPIEN XT THV
Number analyzed (Participants) | 199
percentage of patients | 12.1

2. Secondary Outcome: All Cause Mortality
Time Frame: 30 days
Measure: Number; unit: percentage of patients
Arm/Group | TAVR With SAPIEN XT THV
Number analyzed (Participants) | 199
percentage of patients | 2.5

3. Secondary Outcome: All Cause Mortality
Time Frame: 12 months
Measure: Number; unit: percentage of participants
Arm/Group | TAVR With SAPIEN XT THV
Number analyzed (Participants) | 199
percentage of participants | 8.5

ADVERSE EVENTS:
Time Frame: All-Cause mortality for 12 months of follow-up post-implantation of device, Serious and other Adverse Events for 30-days post-implantation of device are presented.
Description: All Adverse Events are site-reported.
Arm/Group | TAVR With SAPIEN XT THV
All-Cause Mortality (participants affected / at risk) | 17/199
Serious Adverse Events (participants affected / at risk) | 73/199
Other Adverse Events (participants affected / at risk) | 182/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR With SAPIEN XT THV (N=199)
Abnormal lab value (Investigations) | 1 (1)
Access site and access related vascular injury - Dissection (Injury, poisoning and procedural complications) | 4 (4)
Access site and access related vascular injury - Distal embolization (noncerebral) (Injury, poisoning and procedural complications) | 1 (1) — Access site and access related vascular injury - Distal embolization (noncerebral) from vascular source
Access site and access related vascular injury - Failure of percutaneous access site closure (Injury, poisoning and procedural complications) | 2 (2) — Access site and access related vascular injury - Failure of percutaneous access site closure resulting in intervention
Access site and access related vascular injury - Hematoma (Injury, poisoning and procedural complications) | 2 (2)
Access site and access related vascular injury - Pseudoaneurysm (Injury, poisoning and procedural complications) | 3 (3)
Access site and access related vascular injury - Rupture (Injury, poisoning and procedural complications) | 1 (1)
Access site and access related vascular injury - Ventricular rupture (Apical rupture) (Injury, poisoning and procedural complications) | 1 (1)
Anemia/Hemolytic anemia (Metabolism and nutrition disorders) | 4 (4)
Angina/Cardiac chest pain (Cardiac disorders) | 1 (1)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 17 (21)
Bleeding - Hemorrhage (Vascular disorders) | 8 (8)
Cardiac tamponade/Pericardial effusion (Cardiac disorders) | 3 (3)
Device migration/malposition requiring intervention (Injury, poisoning and procedural complications) | 2 (2)
Embolization including air/calcific valve material or Thrombus (Injury, poisoning and procedural complications) | 1 (1)
Gastro Intestinal event - Non-hemorrhagic (Gastrointestinal disorders) | 2 (2)
Heart failure/CHF/Low output failure (Cardiac disorders) | 6 (6)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 7 (7)
Infection - Respiratory infection (Infections and infestations) | 5 (5)
Infection - Urinary tract infection (Infections and infestations) | 2 (2)
Myocardial Infarction (Cardiac disorders) | 2 (2)
Mental state change (not neurological) - Confusion (Psychiatric disorders) | 3 (3)
Miscellaneous - Other (Investigations) | 1 (1)
Multi organ failure (Investigations) | 1 (1)
Neurological - Hemorrhagic stroke (Nervous system disorders) | 1 (1)
Neurological - Ischemic stroke (Nervous system disorders) | 3 (3)
Neurological - Other (Nervous system disorders) | 2 (2)
Neurological - Other new neurological sign consistent with stroke (Nervous system disorders) | 1 (1)
Neurological - TIA (Nervous system disorders) | 1 (1)
Renal insufficiency or renal failure (Renal and urinary disorders) | 4 (4)
Respiratory event - Aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory event - Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Respiratory event - Other (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory event - Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory event - Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Syncope (Vascular disorders) | 3 (3)
Unknown cause of death (Investigations) | 1 (1)
Other (Investigations) | 10 (11)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 2 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TAVR With SAPIEN XT THV (N=199)
Access site and access related vascular injury - Hematoma (Injury, poisoning and procedural complications) | 51 (58)
Anemia/Hemolytic anemia (Metabolism and nutrition disorders) | 21 (21)
Arrhythmia/Conduction system injury (defect) (Cardiac disorders) | 65 (91)
Bleeding - Hemorrhage (Vascular disorders) | 58 (68)
Hypotension (Vascular disorders) | 28 (29)
Musculoskeletal - Pain (Musculoskeletal and connective tissue disorders) | 18 (19)
Other (Investigations) | 100 (160)
Abnormal Labs (Blood and lymphatic system disorders) | 13 (15)
Genito-Urinary event - Non-hemorrhagic (Renal and urinary disorders) | 13 (13)
Hypertension (Cardiac disorders) | 15 (15)
Infection - Respiratory infection (Infections and infestations) | 11 (12)
Mental state change (not neurological) - Confusion (Psychiatric disorders) | 11 (12)
Renal insufficiency or renal failure (Renal and urinary disorders) | 12 (12)
Miscellaneous - Other (General disorders) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No